CLINICAL TRIAL: NCT06211231
Title: MY-ENDO -- Mind Your ENDOmetriosis: a Digital Mindfulness- and Acceptance-based Endometriosis Self-management Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MY-ENDO-digital
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Endometriosis
Keywords: Endometriosis; Quality of life; Digital psychological interventions; Randomized controlled trial; Mindfulness-based intervention; Acceptance and commitment therapy; Pelvic pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of three groups: 1) self-guided digital intervention, 2) therapist-guided digital intervention, or 3) no-treatment control group (waiting list)
Who Masked: Investigator
Masking Description: Only principal investigator is blinded, as neither participants nor care providers can be feasibly blinded, since both parties will know if a video consultation is provided or not. The study includes only patient-reported outcomes, hence, the outcome assessors are the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-guided digital intervention (Experimental): The program consists of 10 online sessions that teach and guide different endometriosis-related themes. The sessions include mindfulness-meditation, yoga, written assignments and patient-education, that are accessed through the digital platform. Participants continue medical treatment as usual.
  Interventions: Behavioral: Digitally delivered mindfulness- and acceptance-based psychological intervention
- Therapist-guided digital intervention (Experimental): The program consists of 10 online sessions that teach and guide different endometriosis-related themes. The sessions include mindfulness-meditation, yoga, written assignments and patient-education, that are accessed through the digital platform. This arm includes 11 online video-consultations with a therapist (one prior to starting and one for each session.) Participants continue medical treatment as usual.
  Interventions: Behavioral: Digitally delivered mindfulness- and acceptance-based psychological intervention
- No-treatment control group (waiting list) (No Intervention): Participants randomized to the waiting list will be offered one of the two experimental treatments. Participants continue medical treatment as usual.

INTERVENTIONS:
Behavioral: Digitally delivered mindfulness- and acceptance-based psychological intervention — MY-ENDO is developed specifically for endometriosis and includes ten themes; one for each session: 1) endometriosis, 2) chronic pain and pain mechanisms, 3) stress, 4) thoughts and feelings, 5) grief, 6) identity and meaning, 7) everyday life and relations, 8) health, diet and exercise, 9) value-based action and 10) a good life with endometriosis.
  Arms: Self-guided digital intervention; Therapist-guided digital intervention

SUMMARY:
The purpose of the study is to assess the effect of a digital mindfulness- and acceptance-based psychological intervention on quality of life, work ability, pain experience and physical and mental health in participants experiencing chronic pain, fatigue and/or reduced quality of life due to endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Signed informed consent.
* Endometriosis diagnosed by a gynecologist based on the medical case history, ultrasound, laparoscopy, or MRI (all self-reported).
* Moderate to severe symptoms (pelvic pain and/or fatigue measured on an 11-point numeric rating scale (NRS) from 0 = no pain/fatigue to 10 = worst imaginable pain/fatigue symptom) or reduced endometriosis-related quality of life (measured by the EHP-30):
* Moderate to severe endometriosis-related chronic pelvic pain (NRS > 2) or
* Moderate to severe endometriosis-related fatigue (NRS > 2) or
* Low endometriosis-related quality of life (one or more EHP-30 subscale mean scores ≥ 40.00).
* Relevant clinical and/or surgical treatment according to the European Society of Human Reproduction and Embryology (ESHRE) guidelines for endometriosis has been attempted.
* Willingness to practice mindfulness and yoga at home for 30-45 minutes 5-7 days a week during the treatment period.

Exclusion Criteria:

* Under 18 years old.
* Severe psychiatric diagnosis made by a psychiatrist and/or ongoing psychiatric treatment.
* Pregnancy or planned pregnancy during the study period.
* An estimated lack of capacity or surplus energy to enter into a digital mindfulness treatment, for instance, because of:
* major life events taking place at the same time (e.g., divorce, loss of a close relative, etc.)
* linguistic or cultural barriers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL) | Change in Endometriosis Health Profile-30 from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization. Primary outcome comparison is between baseline and post-intervention (after session 10.)
  QoL is measured using the Endometriosis Health Profile-30 scale, on a scale from 0 to 100, with higher scores indicating worse quality of life.

SECONDARY OUTCOMES:
Quality of Life subdomains | Change in Quality of Life subdomains from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Quality of Life subdomains will be measured using the six add-on modules to Endometriosis Health Profile-30, on a scale from 0 to 100, with higher scores indicating worse quality of life.
Work ability | Change in Work Ability Index from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Work ability is measured using the Work Ability Index scale, on a scale from 7 to 49, with higher scores indicating better work ability.
Pain and other endometriosis symptoms | Change in pain and other endometriosis symptoms from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Pain and other endometriosis symptoms is measured on numeric rating scales (NRS) ranging from 0 (no pain/no symptom) to 10 (worst pain imaginable/worst symptom imaginable.) Symptoms includes (among others) noncyclical pelvic pain, dysmenorrhea, dysuria, dyspareunia, dyschezia, fatigue, constipation, diarrhea.
Pain acceptance | Change in Chronic Pain Acceptance Questionnaire from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Pain acceptance is measured using the Chronic Pain Acceptance Questionnaire, on a scale from 0 to 120, with higher scores indicating more pain acceptance.
Sleep quality | Change in Pittsburgh Sleep Quality Index from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Sleep quality is measured using the Pittsburgh Sleep Quality Index, on a scale from 0 to 21, with higher scores indicating worse sleep quality.
Fatigue | Change in fatigue from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Fatigue is measured using the Chalder Fatigue Scale, on a scale from 0 to 33, with higher scores indicating more fatigue.
Wellbeing | Change in World Health Organization - Five Wellbeing Index from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Wellbeing is measured using the World Health Organization - Five Wellbeing Index, on a scale from 0 to 25, with higher scores indicating better wellbeing.
Pain catastrophizing | Change in Pain Catastrophizing Scale from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Pain catastrophizing is measured using the Pain Catastrophizing Scale, on a scale from 0 to 52, with higher scores indicating more severe pain catastrophizing.
Anxiety symptoms | Change in Generalized Anxiety Disorder Screener from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Anxiety symptoms will be measured using the Generalized Anxiety Disorder Screener, on a scale from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Depressive symptoms | Change in Beck's Depression Inventory from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Depressive symptoms will be measured by Beck´s Depression Inventory, on a scale from 0 to 63, with higher scores indicating more severe depressive symptoms.
Perceived stress | Change in Perceived Stress Scale from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Perceived stress will be measured by The Perceived Stress Scale, on a scale from 0 to 40, with higher scores indicating higher perceived stress.
Psychological flexibility | Change in Acceptance and Action Questionnaire-II from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Psychological flexibility will be measured by the Acceptance and Action Questionnaire-II (AAQ-II), on a scale from 7 to 49, with higher scores indicating less psychological flexibility.
Mindfulness | Change in Five Facet Mindfulness Questionnaire from pre-randomization to after sessions 5 and 10, and 3, 6 and 12 months post-randomization.
  Mindfulness will be measured by the Five Facet Mindfulness Questionnaire, on a scale from 39 to 195, with higher scores indicating more mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Marschall, MSc, Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Department of Gynaecology and Obstetrics, Aarhus, Central Jutland
  - The Danish Endometriosis Patients Association, Billund

IPD SHARING:
Plan to Share IPD: Yes
When participant inclusion has ended, data can be shared in accordance with the International Committee of Medical Journal Editors (ICJME) guidelines, if relevant research objectives are provided. Data sharing will require approval from the Research Ethics Committee in Denmark and the Danish Data Protection Agency, and the requesting party shall cover any fees associated with data sharing. Requests for data can be addressed to hmars@psy.au.dk.